CLINICAL TRIAL: NCT05694897
Title: Ultrasound Guided Erector Spinae Block Using a Combination of Bupivacaine and Dexmedetomidine Versus Bupivacaine and Magnesium Sulfate for Postoperative Analgesia in Lumbar Spine Surgery
Brief Title: Erector Spinae Block Using a Dexmedetomidine Versus Magnesium Sulfate as an Adjuvant to Bupivacaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sameh Refaat, Lecturer of anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M d 538/2020
Record Dates: First submitted 2022-12-24; First posted 2023-01-23 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Analgesia
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae block using a combination of bupivacaine and magnesium sulfate (Active Comparator): Ultrasound guided erector spinae block at the level of T10 using a combination of 20 ml bupivacaine 0.25% and 3.75ml magnesium sulfate for treatment of postoperative pain
  Interventions: Procedure: Erector spinae block using bupivacaine 0.25% and magnesium sulfate
- Erector spinae block using a combination of bupivacaine and dexmedetomidine (Active Comparator): Ultrasound guided erector spinae block at the level of T10 using a combination of 20 ml bupivacaine 0.25% and 1ug/kg dexmedetomidine for treatment of postoperative pain
  Interventions: Procedure: Erector spinae block using bupivacaine and dememdetomidine

INTERVENTIONS:
Procedure: Erector spinae block using bupivacaine 0.25% and magnesium sulfate — After induction of general anesthesia the patients will be flipped to the prone position and ESP block was performed using, a high frequency linear ultrasound probe placed longitudinally 2 to 3 cm lateral to the 10th thoracic vertebrae, and the trapezius and erector Spinae muscles identified.
  An 18-G Tuohy needle passed along the plane of the transducer until its tip hit the transverse process of T10; the needle was then withdrawn slightly.
  Total volume of 25 ml was injected including 20 mL 0.25% bupivacaine plus 3.75 ml NS and 125 mg MgSO4 (1.25ml).
  Arms: Erector spinae block using a combination of bupivacaine and magnesium sulfate
Procedure: Erector spinae block using bupivacaine and dememdetomidine — After induction of general anesthesia the patients will be flipped to the prone position and ESP block was performed using, a high frequency linear ultrasound probe placed longitudinally 2 to 3 cm lateral to the 10th thoracic vertebrae, and the trapezius and erector Spinae muscles identified.
  An 18-G Tuohy needle passed along the plane of the transducer until its tip hit the transverse process of T10; the needle was then withdrawn slightly.
  Total volume of 25 ml was injected including 20 mL 0.25% bupivacaine plus dexmedetomidine 1ug/kg.
  Arms: Erector spinae block using a combination of bupivacaine and dexmedetomidine

SUMMARY:
This prospective parallel group randomized study will be conducted over 52 adult participants between 20 and 60 years ASA (American Association of Anesthesiologists) I and II undergoing lumbar spine surgery. The participants will be randomly allocated into 2 groups. Group BM (Bupivacaine + magnesium sulfate) will receive bilateral erector spinae block using bupivacaine and magnesium sulfate after induction of general anesthesia, while group BD (Bupivacaine + dexmedetomidine) will receive bilateral erector spinae block using bupivacaine and dexmedetomidine after induction of general anesthesia. Hemodynamic changes will be monitored intraoperatively, and postoperative pain will be assessed using the visual analogue scale in order to assess the need for postoperative analgesia.

DETAILED DESCRIPTION:
This prospective parallel group randomized study will be conducted over 52 adult participants between 20 and 60 years ASA (American Association of Anesthesiologists) I and II undergoing lumbar spine surgery. The participants will be randomly allocated into 2 groups.

General anesthesia will be induced using propofol 1-2mg/kg, fentanyl 2ug/kg, and atracurium 0.5mg/kg.

Both groups will receive bilateral erector spinae block Group BM will receive bilateral erector spinae block .A technique that will be performed ultrasound guided to identify the transverse process of T10, and an 18G (gauge) needle will be introduced in plane deep to the erector spinae muscle after which a combination of 20ml bupivacaine 0.25% and 2.5 ml magnesium sulfate.

While group BD will receive the same block with the with 20ml bupivacaine 0.25% and dexmedetomidine 1ug/kg.

Hemodynamic changes will be monitored intraoperatively, for detection of any variations.

Postoperative pain will be assessed every 2 hours following the surgery using the visual analog scale in order to assess the need for postoperative analgesia.

Analgesia will be given in the form of nalbuphine 10mg when the visual analog scale is above 4.

Patient satisfaction will be measured by a scale from 1-10 the next day. Any complications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1, and 2

Exclusion Criteria:

* Patient refusal
* Spine deformities
* Coagulopathies
* Infection at the site of surgery
* Body weight above 100kg
* Known allergy to used drugs
* Psychiatric illness

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Measurement of the duration of postoperative analgesia | 12 hours
  Postoperative analgesia duration will be assessed using the visual analogue scale which is from 0-10 were 0 means no pain and 10 is the worst pain
Dose of postoperative nalbuphine | 12 hours
  Total dose of postoperative nalbuphine will be measured depending on the visual analogue scale

SECONDARY OUTCOMES:
Patient satisfaction | 48 hours
  Patient satisfaction will be measured using the patient satisfaction scale which will be from 1-10 were 1 means no satisfaction and 10 is the best satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided